CLINICAL TRIAL: NCT03780361
Title: Changes in Inflammatory Biomarkers Including Soluble CD14 and Hyperreflective Foci in Diabetic Macular Edema Patients Treated With Aflibercept (FORESIGHT)
Brief Title: Changes in Inflammatory Biomarkers Including Soluble CD14 and Hyperreflective Foci in DME Patients Treated With Aflibercept (FORESIGHT)
Acronym: FORESIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hyewon Chung (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Hyewon Chung, Associate professor, Konkuk University Medical Center
Organization: Konkuk University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20658
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Macular Edema
Keywords: soluble CD14; MCP-1; IL-6; ICAM-1; cytokine; visual acuity; optical coherence tomography; macular thickness; hyperreflective foci
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aflibercept injection group (Experimental): drug: Eylea (aflibercept) (11.12mg/0.278ml) dose: 2mg (0.05ml) usage: With topical anesthesia and intravitreal injection of aflibercpt in aseptic condition.
  frequency and duration: monthly intravitreal aflibercept injections.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Total 5 times of monthly intravitreal aflibercept injections will be done.
  Other Names: Eylea

SUMMARY:
This study evaluates the effect of aflibercept on the change of cytokines incluing sCD14, MCP-1, IL-6, and ICAM-1 in the aqueous humor of DME patients. Additionally, changes of visual acuity (ETDRS), optical coherence tomography parameters including hyperreflective foci and thickness of macula are also investigated.

DETAILED DESCRIPTION:
Intraocular steroid agents have been shown to decrease inflammatory cytokines in diabetic macular edema (DME) patients and thus have roles in the treatment of these patients. However, I believe that anti-VEGF could effectively decrease intraocular inflammatory responses in these patients with much fewer side effects than intraocular steroid agents.

Since soluble CD14 (sCD14) is the known marker of inflammatory cells including microglia, increased or decreased retinal inflammation accompanied by DME could be monitored using sCD14 in patients with DME. Recently, I published an article regarding the strong association of increased sCD14 in the aqueous humor (AH) from DME patients, especially in increased inner retinal edema as well as increased hyper reflective foci (HF) in optical coherence tomography (OCT). This associated changes of sCD14 levels and HF in the retina suggested that the HF might represent the activated microglia in DME. I also showed that the intravitreal bevacizumab injection resulted in a reduction of sCD14 in the AH and HF in OCT. However, that study was retrospective and I could not have many patients' follow-up data after bevacizumab treatments and thus was not able to get conclusive results regarding decreased retinal inflammation after anti-VEGF. Therefore, I believe that a well-desinged prospective study is needed to clarify whether retinal inflammation is ameliorated after anti-VEGF treatment. Moreover, I believe that aflibercept is more appropriate and better drug than bevacizumab to investigate the changes in the cytokine levels along with the improvement of inflammatory milieu in DME due to the following reasons. First, recent DRCR.net Protocol-T reported the superior clinical outome of aflibercept compared to bevacizumab on DME. Second, aflibercept has significantly higher binding affinity to VEGF-A compared to ranibizumab or bevacizumab. Third, aflibercept also binds to VEGF-B and placental growth factor (PlGF), unlike ranibizumab or bevacizumab. PlGF-VEGFR1 pathway contributes to inflammation by triggering production of proinflammatory cytokines.

Thus, I would like to investigate the efficacy of aflibercept for reducing inflammation in DME. Therapeutic effects of aflibercept on reduction of DME in the context of amelioration of inflammation will be proved using sCD14 and HF as surrogate markers in this proposed study. Besides sCD14, tracking the cytokines including MCP-1, IL-6, and ICAM-1 in the AH in a well-controlled prospective setting of aflibercept treatments will enhance our understanding regarding the role of inflammation on DME, and the importance of aflibercept for decreasing ocular inflammation in DME patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 19 years with type 1 or 2 diabetes mellitus.
2. Patients with DME secondary to diabetes mellitus involving the center of the macula (defined as the OCT center subfield) in the study eye.
3. Decrease in vision determined to be primarily the result of DME in the study eye.
4. BCVA ETDRS letter score of 80 to 24 (20/25 to 20/320) in the study eye.
5. Retinal thickness ≥ 300 µm as assessed by OCT in the study eye.
6. Willing and able to comply with clinic visits and study-related procedures.

Exclusion Criteria:

1. Ocular conditions with a poorer prognosis in the fellow eye than in the study eye.
2. History of vitreoretinal surgery in the study eye.
3. Previous treatment with intraocular anti-angiogenic drugs (bevacizumab, ranibizumab etc.) or laser photocoagulation in the study eye within 90 days.
4. Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of day 1.
5. Invasive intraocular surgery incluing cataract surgery within 90 days of day 1.
6. Yttrium-aluminium-garnet capsulotomy in the study eye within 30 days before day 1.
7. Aphakia in the study eye.
8. Vitreomacular traction or epiretinal membrane in the study eye evident on OCT that is thought to affect central vision.
9. Active proliferative diabetic retinopathy in the study eye.
10. Current iris neovascularization in the study eye.
11. Evidence of infection including infectious blepharitis, keratitis, scleritis, conjunctivitis or endophthalmitis in either eye.
12. Uncontrolled glaucoma in the study eye or filtration surgery for glaucoma in the past or likely to be needed in the future on the study eye.
13. Intraocular pressure ≥25 mmHg in the study eye.
14. Myopia of a spherical equivalent prior to any possible refractive or cataract surgery of ≥ -8 diopters.
15. Concurrent disease in the study eye, other than DME, that could compromise VA, require medical or surgical intervention during the study period, or could confound interpretation of the results (including uveitis, retinal vascular occlusion, retinal detachment, macular hole, significanlty large hard exudate at macula, atrophy of retinal pigment epithelium, submacular scar, macular isdhemia, or choroidal neovascularization).
16. Only one functional eye even if that eye is otherwise eligible for the study.
17. Ocular media of insufficient quality to obtain fundus and OCT images.
18. Current treatment for a serious systemic infection.
19. Administration of systemic anti-angiogenic agents within 180 days before day 1.
20. Pregnant women, pregnancy planning during the study period, lactating
21. Severe active intraocular inflammation is observed in the eyes injected with Aflibercept
22. History of hypersensitivity to Aflibercept or excipient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the level of sCD14 in the aqueous humor | From baseline to week 20
  Change in the level of sCD14 in the aqueous humor measured by ELISA

SECONDARY OUTCOMES:
Change in the levels of cytokines (MCP-1, IL-6, ICAM-1) in the aqueous humor | From baseline to week 20
  Change in the levels of cytokines (MCP-1, IL-6, ICAM-1) in the aqueous humor measured by ELISA
Change in the number of hyperreflective foci (HF) on optical coherence tomography (OCT) | From baseline to week 20
  Change in the number of HF on optical coherence tomography OCT B-scan
Change in the thickeness of macula on OCT | From baseline to week 20
  Change in the thickeness of macula on OCT
Change in mean visual acuity (ETDRS) | From baseline to week 20
  Change in mean visual acuity (ETDRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee H, Jang H, Choi YA, Kim HC, Chung H. Association Between Soluble CD14 in the Aqueous Humor and Hyperreflective Foci on Optical Coherence Tomography in Patients With Diabetic Macular Edema. Invest Ophthalmol Vis Sci. 2018 Feb 1;59(2):715-721. doi: 10.1167/iovs.17-23042. PMID 29392317